CLINICAL TRIAL: NCT05431751
Title: Clinical Proof-of-concept Study on Immune Surveillance and Alertness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 153-012
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2022-08

CONDITIONS: Immune Surveillance

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, cross-over study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group A (Experimental): Crossover study: Participants will be consuming placebo on a clinic day at least 1 week prior to a clinic day where they will consume the active intervention. Following the second clinic day, the participant will consume active intervention for 7 days. The participant will then undergo a washout period of 7 days.
  Interventions: Dietary Supplement: Whole Algae

INTERVENTIONS:
Dietary Supplement: Whole Algae — Whole Euglena gracilis algae, produced by proprietary fermentation.

SUMMARY:
Clinical proof-of-concept study comparing the acute. effects of an algae-based dietary supplement on immune surveillance and alertness. This study involves twenty-four participants composed of healthy adults, who will be taking either a placebo or supplement at different times. Testing for immune status, cytokine levels, and immune responsiveness will be conducted to determine the acute impact of the supplement on immune function compared to a placebo.

Long term effects and lingering effects will be tested using the same parameters, following a consumption period of one week, as well as a washout period of one week.

DETAILED DESCRIPTION:
Clinical-proof-of-concept study comparing the acute immune effects as well as the lasting and lingering effects of a dietary supplement, and a placebo. The dietary supplement is composed of whole Euglena gracilis algae, produced using a proprietary fermentation technique.

24 subjects will participate in a placebo-controlled, double-blinded, cross-over study design, wherein they will be taking placebo, or dietary supplement each separated by a 1-week washout period to evaluate rapid effects. Following which the subjects will also be taking placebo or dietary supplement continuously for 1 week each, to evaluate the long term and lingering effects.

For acute evaluation, blood samples are taken 1 hour after participants arrive, the dose is then administered. Samples are take 1 hour and 2 hours following administration. For long-term and lingering evaluation, blood samples are taken 1 hour after participants arrive. At all blood sample collections, a spit sample will also be taken for salivary IgA testing.

A series of immune panels will be used to determine the acute impacts on immune surveillance, immune cell activation status, immune cell priming, and cytokine profiles. Ex vivo immune challenges and salivary IgA testing will be used to determine the direct impacts on immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Veins easy to see in both arms
* Willing to comply with a 24-hours wash-out period for vitamins and nutritional supplements
* Willing to comply with study procedures, including maintaining a consistent diet and lifestyle routine throughout the study. Consistent habit of bland breakfasts on days of clinic visits, abstaining from exercising, tobacco use, and nutritional supplements on the morning of a study visit, abstaining from use of coffee, tea, and soft-drinks for at least one hour prior to a clinic visit
* Willing to abstain from music, candy, gum, computer/cellphone use during clinic visits

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder)
* Taking anti-inflammatory medications on a daily basis (81 mg aspirin is acceptable)
* Vaccination during past 2 weeks
* Currently experiencing intense stressful events/ life changes
* Currently in intensive athletic training (such as marathon runners)
* Currently taking antipsychotic medications such as clozapine, Risperdal, Abilify, Zyprexa or Seroquel
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights)
* Unwilling to maintain a constant intake of supplements over the duration of the study
* Anxiety about having blood drawn
* People of childbearing potential: Pregnant, nursing, or trying to become pregnant
* Known food allergies or sensitivities related to the test product or placebo
* Prescription medication will be evaluated on a case-by-case basis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Immune Surveillance and Alerness | 2 hours, 1 week
  Observation of changes in immune cell trafficking and status of immune cell alertness, ie. the changes in immune cell populations and activation following administration.

SECONDARY OUTCOMES:
Immune communication | 2 hours, 1 week
  Observation of changes in serum cytokine levels

OTHER OUTCOMES:
Immune Responsiveness | 2 hours, 1 week
  Ex vivo immune challenges, observing the capabilities of anti-bacterial and anti-viral defenses. Additionally, mucosal immune protection as determined by salivary IgA, defensins, and transferrin changes .

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No